CLINICAL TRIAL: NCT07271095
Title: Strengthening Numerical Skills and Medication Calculation Abilities of Nursing Students Through Peer Education: A Randomized Controlled Trial
Brief Title: Strengthening Numerical Skills and Medication Calculation Abilities of Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lokman Hekim University (Other Government)
Responsible Party: Principal Investigator, Beratiye Oner, Assistant Professor, Lokman Hekim University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024146
Record Dates: First submitted 2025-11-25; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Student; Nursing
Keywords: Nursing education; peer education; Medication calculation; Numerical skills

STUDY DESIGN:
Intervention Model Description: This study employed a randomized controlled pretest-posttest experimental design to evaluate the effectiveness of peer-assisted education on nursing students' numerical and drug calculation skills. Participants were randomly assigned to either the experimental group (n=27) or the control group (n=28). The intervention model consisted of a three-week peer-assisted training program comprising five structured sessions. Each session was conducted by trained mentor students who facilitated small group learning activities. During the sessions, students collaboratively solved numerical and drug calculation problems, discussed solution strategies, and received formative feedback from peers and mentors. The control group continued with the standard nursing curriculum without peer support. This interventional model was designed to foster active learning, peer collaboration, and problem-based engagement, aiming to enhance students' cognitive and practical competencies in medication calculation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Peer-supported medication calculation training program
  Interventions: Other: Peer-supported medication calculation training
- Control Group (No Intervention): Participants who received traditional lecture-based instruction

INTERVENTIONS:
Other: Peer-supported medication calculation training — The intervention consisted of a peer-supported education program on medication dosage calculation, implemented over three weeks with five 60-minute sessions. In Week 1, four mentor students-senior nursing students with prior training in medication calculations and a GPA above 3.0-received refresher instruction from the course instructor. The training covered decimals, percentages, unit conversions, weight-based and non-weight-based dose calculations, and infusion pump adjustments, followed by sample problem-solving activities. The intervention group was divided into four subgroups, each consisting of 7-8 students, and each was assigned a consistent mentor. Each session included 30 minutes of individual and peer problem-solving followed by 30 minutes of guided mentoring. The course instructor provided supervision and feedback throughout the sessions. During Weeks 2 and 3, students practiced numerical and medication dosage calculations through peer-supported exercises.
  Arms: Intervention Group

SUMMARY:
This experimental study aims to evaluate the effect of peer-assisted education on nursing students' numerical and drug calculation skills. A randomized controlled pretest-posttest design will be conducted with 55 first-year nursing students (27 in the experimental group and 28 in the control group). The experimental group will participate in a three-week peer education program focusing on numerical problem-solving and medication dosage calculations, led by trained mentor students.

ELIGIBILITY:
Inclusion Criteria:

* Students who were registered for the Fundamentals of Nursing course for the first time
* Students who agreed to participate in the research voluntarily

Exclusion Criteria:

* Students who graduated from a Health Vocational High School
* Students who had previous training in the health field
* Students who had previously taken a Fundamentals of Nursing course
* Students diagnosed with a psychiatric illness
* Students who were regularly taking psychiatric medications
* Students who did not attend the theoretical sessions of the course

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
The Medication Calculation Ability | They were evaluated before the intervention and after 3 weeks of intervention.
  Medication Calculation Ability Assessment Form (Pre-Test, Post-Test): The pre-test consisted of eight questions. The posttest consisted of twenty questions, including additional questions similar to those in the pretest. The questions covered the following categories:
  * Dosage calculation for solid and liquid oral medications (3 questions in the pretest, 8 questions in the posttest),
  * Dosage calculation for injections (3 questions in the pretest, 7 questions in the posttest),
  * Calculation of percentage solutions and intravenous fluids (2 questions in the pretest, 5 questions in the posttest).
  Each correct answer was scored; the participants' correct answers were averaged to convert the score into a percentage. Thus, a medication calculation skill score ranging from 0% to 100% was obtained for each participant.

SECONDARY OUTCOMES:
The Numerical Skills | They were evaluated both before and after the 3-week intervention.
  Numerical Skills Assessment Form (Pre-Test, Post-Test): The pre-test consisted of five questions. The post-test consisted of 10 questions, including additional questions similar to those in the pre-test. The questions covered basic numerical skills, including addition, subtraction, multiplication, division, fractions, decimals, percentage calculations, and unit conversions. Each correct answer was scored, and the percentage score was converted by averaging the number of correct answers. Thus, a numerical skill score ranging from 0% to 100% was obtained for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Beratiye Oner, Study Director — Lokman Hekim University
Locations (1):
- Lokman Hekim University, Çankaya, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No